CLINICAL TRIAL: NCT01866176
Title: Effects of a New Knee Brace for Treatment of the Knee Osteoarthritis on the Medial Knee Loading During Gait
Brief Title: Effects of a New Knee Brace for Treatment of the Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Fonds de la Recherche en Santé du Québec (Other Government); Ergorecherche Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OG2007-097-A4
Record Dates: First submitted 2013-05-09; First posted 2013-05-31 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Knee osteoarthritis patients (Experimental): Knee osteoarthritis patients with Kellgren & Lawrence grade I, II or III Stabilizing Knee Brace Valgus Knee Brace New Knee Brace
  Interventions: Device: Stabilizing Knee Brace; Device: Valgus Knee Brace; Device: New Knee Brace

INTERVENTIONS:
Device: Stabilizing Knee Brace — Brace with no valgus action
Device: Valgus Knee Brace — Valgus brace with traditional three point bending system
Device: New Knee Brace — Brace with new mechanism to decrease the knee loading.

SUMMARY:
The purpose of this study is to evaluate the immediate effects of a knee brace with a new mechanism on the pain and medial knee loading during gait among medial knee osteoarthritis patients. The effects of this new brace is compared to a stabilizing brace and a typical valgus knee brace. The investigators recruited 24 knee osteoarthritis and they have to wear each of the three braces during three months. A fifteen days wash-out period is given after each three months. Biomechanical evaluation is carried out before and after each three months. This evaluation consisted of three questionnaires (KOOS, WOMAC and Medical Outcome Score Short Form-36 (MOS-SF36)), a motion analysis with an optoelectronic system, then a 6-min walk test. During motion analysis, ten gait trials are executed without brace and ten with the brace.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic medial knee OA (Kellgren-Lawrence grade I, II or III) according to clinical and radiological criteria of the American College of Rheumatology
* Knee pain > 31/100 (Western Ontario and McMaster Universities Arthritis Index - WOMAC)
* Moderately active
* Varus knee alignment equal or superior to 2°

Exclusion Criteria:

* Severe knee OA (K-L grade IV)
* Rheumatoid arthritis or other inflammatory arthritis
* Avascular necrosis
* History of periarticular fracture or septic arthritis
* Bone metabolic disease
* Pigmented villonodular synovitis
* Cartilaginous disease
* Neuropathic arthropathy
* Synovial osteochondromatosis
* Total or partial knee arthroplasty
* Flexion contracture of ipsi- or contra-lateral knee greater than 15°
* Hip or ankle joint damage with mobility limitation
* Obesity (BMI ≥ 40)
* Intra-articular corticosteroids injection in the affected knee during the two previous months
* Reduced mobility (Charnley class C)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Knee adduction moment | Change from Baseline at 3 months
Change in Knee pain | Change from Baseline at 3 months
  A 20-cm visual analog scale (0-100) is used to assess pain.

SECONDARY OUTCOMES:
Change in Spatiotemporal gait parameters | Change from Baseline at 3 months
  Test of the gait symmetry with the gait phase duration and step length.
Change in Gait velocity | Change from Baseline at 3 months
Change in Knee adduction angle | Change from Baseline at 3 months
Change in Knee brace comfort | Change from Baseline at 3 months
  A 20-cm visual analog scale (0-100) is used to assess comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Corbeil, PhD, Study Director — Laval University; Yoann Dessery, MSc, Principal Investigator — Laval University; Étienne L Belzile, MD, Study Director — Laval University
Locations (1):
- Pavillon de l'Éducation Physique et des Sports - Université Laval, Québec, Quebec, Canada